CLINICAL TRIAL: NCT05017675
Title: Comparing the Effect of a High SFA Diet and High Fructose Diet on Hepatic Insulin Sensitivity
Brief Title: Effect of Dietary SFA and Fructose on Hepatic Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NL78281.068.21
Record Dates: First submitted 2021-08-10; First posted 2021-08-24 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Insulin Resistance
Keywords: High fructose diet; High saturated fat diet; De novo lipogenesis; Hepatic saturated fatty acids
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High fructose diet (Experimental): Participants will receive dietary products high in fructose for 4 weeks.
  Interventions: Other: High fructose diet
- High saturated fat diet (Experimental): Participants will receive dietary products high in saturated fat for 4 weeks.
  Interventions: Other: High saturated fat diet

INTERVENTIONS:
Other: High fructose diet — 4 week high fructose diet.
  Intended composition (En%):
  Carbohydrates: 60-70 Fat: 20-30 Protein: 10-15 Fructose: 20 SFA: 5
  Arms: High fructose diet
Other: High saturated fat diet — 4 week high saturated fat diet.
  Intended composition (En%):
  Carbohydrates: 35-45 Fat: 40-50 Protein: 10-15 Fructose: 5 SFA: 20
  Arms: High saturated fat diet

SUMMARY:
High rates of de novo lipogenesis (DNL) and high saturated fatty acid (SFA) fraction in the liver both have been associated with poor metabolic health and hepatic insulin resistance. Interestingly, the end product of DNL is mainly SFA. So far it is unknown whether it is the process of DNL or the accumulation of SFA per se that leads to hepatic insulin resistance. Therefore, it is of interest to compare the effect of a diet that modifies directly hepatic SFA content (4-week high SFA diet) and a diet that changes SFA indirectly by modifying rates of DNL (4-week high fructose diet). To this end, 18 overweight/obese, but otherwise healthy, males and females will take part in the randomized dietary interventions. The primary outcome is hepatic insulin sensitivity (suppression of EGP during clamp) upon a 4-week high SFA diet versus a 4-week fructose diet.

DETAILED DESCRIPTION:
Rationale: High rates of de novo lipogenesis (DNL) and high saturated fatty acid (SFA) fraction in the liver both have been associated with poor metabolic health and hepatic insulin resistance. Interestingly, the end product of DNL is mainly SFA. So far it is unknown whether it is the process of DNL or the accumulation of SFA per se that leads to hepatic insulin resistance. This is a clinically relevant question, as it will give novel insights towards the best strategy for prevention and treatment of hepatic insulin resistance. Therefore, it is of interest to compare the effect of a diet that modifies directly hepatic SFA content (high SFA diet) and a diet that changes SFA indirectly by modifying rates of DNL (high fructose diet).

Objective: To determine the effect of a 4-week high SFA diet compared to a 4-week high fructose diet on hepatic insulin sensitivity, on hepatic SFA fraction and DNL.

Study design: This is a randomized intervention study comparing the effects of a 4-week high SFA diet compared to a 4-week high fructose diet on hepatic insulin sensitivity.

Study population: 24 overweight/obese, but otherwise healthy, males and females (BMI 27-38 kg/m2), 45-75 years, will participate in the study. Of these 24 included participants, 18 are expected to meet the study criteria and take part in the measurements following the screening, of these 14 need to complete the study.

Intervention: Participants follow a 4-week high SFA diet and a 4-week high fructose diet.

Main study parameters/endpoints: The primary outcome is hepatic insulin sensitivity (suppression of EGP during clamp) upon a 4-week high SFA diet versus a 4-week fructose diet. Secondary outcomes are DNL upon 4-week high SFA versus 4-week high fructose, and delta (baseline-end intervention) hepatic SFA fraction upon 4-week high SFA versus 4-week high fructose.

ELIGIBILITY:
Inclusion Criteria:

* Participants are able to provide signed and dated written informed consent prior to any study specific procedures
* Participants should have suitable veins for cannulation or repeated venipuncture
* Women are post-menopausal (defined as at least 1 year post cessation of menses)
* Aged ≥ 45 and ≤ 75 years
* Body mass index (BMI) 27 - 38 kg/m2
* Stable dietary habits (no weight loss or gain >5kg in the past 3 months)
* Sedentary lifestyle (not more than 2 hours of sports per week)
* No signs of active cardiovascular disease, liver or kidney malfunction
* Liver fat content ≥ 2% weight/weight.

Exclusion Criteria:

* Type 2 diabetes
* Previous enrolment in a clinical study with an investigational product during the last 3 months or as judged by the Investigator
* Patients with congestive heart failure and and/or severe renal and or liver insufficiency or another condition that may interfere with outcomes measured in this study.
* Any contra-indication MRI scanning
* Alcohol consumption of >2 servings per day for men and >1 servings per day for woman
* Smoking in the past 6 months
* Men: Hb <8.4 mmol/L, Women: Hb <7.8 mmol/l
* Vegetarian, vegan, food intolerant to common foods (e.g. gluten intolerant, lactose intolerant)
* Medication use that may influence outcome parameters

A medical doctor will judge participation eligibility based on the medical history questionnaire, medication use and fasting blood parameters. If the medical doctor advises that a volunteer cannot participate, the volunteer will be excluded from enrollment.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Hepatic insulin sensitivity measured by hyperinsulinemic-euglycemic clamp. | after 28 days of each diet
  difference in EGP suppression after the high SFA diet and the high fructose diet

SECONDARY OUTCOMES:
Hepatic fat composition measured by proton magnetic resonance spectroscopy | first day of each diet - after 28 days of each diet
  The change in liver fat composition (%SFA, %MUFA and %PUFA) after the high SFA diet and the high fructose diet
De novo lipogenesis measured by deuterated water | after 25 days of each diet
  Difference between overnight DNL after the high SFA diet and the high fructose diet. Measured as relative contribution of newly synthesized palmitate in the VLDL-TG pool expressed as %DNL.

OTHER OUTCOMES:
Liver fat content measured by proton magnetic resonance spectroscopy | after 28 days of each diet
  Difference in liver fat content after the high SFA diet and the high fructose diet
Peripheral and whole-body Insulin sensitivity measured by hyperinsulinemic-euglycemic clamp | after 28 days of each diet
  Whole body insulin sensitivity is measured as GIR in μmol/kg/min and peripheral insulin sensitivity is measured as Rd in μmol/kg/min. Difference in GIR and Rd after the high SFA diet and the high fructose diet will be determined
Fat oxidation measured by indirect calorimetry | after 25 and 28 days of each diet
  Fat oxidation as determined by indirect calorimetry, will be compared between the high SFA and high fructose diet
Carbohydrate oxidation measured by indirect calorimetry | after 25 and 28 days of each diet
  Carbohydrate oxidation as determined by indirect calorimetry will be compared between the high SFA and high fructose diet
Sleeping metabolic rate measured by indirect calorimetry | after 25 days of each diet
  Sleeping metabolic rate as determined by indirect calorimetry will be compared between the high SFA and high fructose diet
Body composition measured by BodPod | day 1
  Body composition is measured using the BodPod technique and percentage fat mass will be determined for participant characterization.

CONTACTS AND LOCATIONS:
Overall Officials: Vera Schrauwen-Hinderling, Dr, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No
Data can be obtained with the principal investigator if desired.